CLINICAL TRIAL: NCT06166784
Title: Cinical Outcomes of Mectascrew B Interference Screw
Brief Title: Interference Screw Mectascrew-B Postmarket Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P07.001.08
Record Dates: First submitted 2023-11-30; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Injuries Posterior Cruciate Ligament Tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Mectascrew B
  Interventions: Device: Mectascrew B

INTERVENTIONS:
Device: Mectascrew B — reconstruction of ACL or PCL rupture

SUMMARY:
An observational prospective study with the aim to assess the clinical outcomes at 1year after surgery for a specific composite IS (Medacta Mectascrew B) in the reconstructive treatment of ruptured ACL or PCL by means of an autograft or allograft.

DETAILED DESCRIPTION:
This is an observational prospective study with the aim toassess the clinical outcomes at 1year after surgery for a specific composite IS (Medacta Mectascrew B) at 12 months following ACL or PCL reconstruction.

Patients with an ACL or PCL tear scheduled for surgery at OCM Klnik GmbH hospital will be enrolled in the study, after the subscription of informed consent.

The injured ligament will be restored with an auto- or allograft that will be fixed with a composite IS (Mectascrew-B, Medacta International SA). Data concerning demography, preoperative clinical conditions, surgical details including device implanted, tendon harvesting procedure and complications occurred, postoperative clinical data (as per standard practice at 6 weeks, 6 and/or 12 months) will be prospectively collected, in order to assess the functional outcomes (IKDC objective and subjective) and the knee stability (ROM, Pivot Shift or Reverse Pivot Shift test, anterior or posterior drawer test) of the patients.

The treated knee will be also evaluated radiologically by std x-ray according to standard practice to assess swelling, tunnel widening, and resorption problems. The results of this exam will be correlated to the pre-operative findings and to the functional and clinical outcomes evaluated with the different forms

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Patients older than 18 years
* ACL or PCL damage requiring primary ACL or PCL reconstruction
* Patient requiring ACL or PCL surgery with the use of Medacta MectaScrew B interference screw, according to Manufacturer IFU's, i.e. reconstructive therapy of ruptures to the anterior or posterior cruciate ligament by means of autologous grafts
* Patients who are willing to participate in the study and have signed informed consent form.

Exclusion Criteria:

* Patients with contraindications according to IFU's
* Patients with malignant diseases (at the time of surgery)
* Patients with proven or suspected infections (at the time of surgery)
* Patients with functional deficits on the affected extremity (at the time of surgery)
* Patients with known incompatibility or allergy to products materials (at the time of surgery)
* Concomitant ligament injury (grade ≥ 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with an ACL or PCL rupture, and meeting the inclusion/ exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes evaluation | 12 months
  Assessment throught IKCD score. a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

SECONDARY OUTCOMES:
Mobility outcomes evaluation | 6 weeks, 6 months, 12 months
  Assessment throught Range Of Motion of operated knee calculated as degree
Knee stability evaluation of ACL intervention | 6 weeks, 6 months, 12 months
  Pivot shift test. A positive test indicate an injury at ACL
ACL integrity assessment | 6 weeks, 6 months, 12 months
  Anterior drawer test. An anterior translation more than 6 mm indicate a positive test with injuried ACL
Knee stability evaluation of PCL intervention | 6 weeks, 6 months, 12 months
  Reverse Pivot Shift test. In the presence of a posterolateral injury with the knee flexed, the tibia follows gravity and drops into posterolateral subluxation (positive Reverse Pivot Shift Test).
PCL integrity assessment | 6 weeks, 6 months, 12 months
  Posterior drawer test. The test is considered positive if there is a lack of end feel or excessive posterior translation
Interference screw integration | 6 weeks, 6 months, 12 months
  Evaluation of ligament osteointegration, femoral/tibial tunnel widening, presence of fluid in the femoral/tibial tunnel by std x-ray
Incidence of adverse event | 6 weeks, 6 months, 12 months
  collection of adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- OCM Klinik GmbH, Münich, Germany

IPD SHARING:
Plan to Share IPD: No